CLINICAL TRIAL: NCT05278650
Title: Senior PharmAssist: Co-Design and Evaluation of a Toolkit to Promote Scalable Implementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00110307
Record Dates: First submitted 2022-03-04; First posted 2022-03-14 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Medication Therapy Management; Implementation Science

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Communities Adopting Senior PharmAssist Implementation Toolkit (Other): Three communities will commit to learning how to implement the evidence-based, multi-component intervention, Senior PharmAssistTM (SPA), designed to improve function and quality of life of older adults with limited incomes using the SPA toolkit.
  The toolkit, co-developed with community leaders, will help to create a community model for implementation that addresses equitable access to medications, medication management, and community supports that promote physical function and healthy aging in place.
  Interventions: Other: Senior PharmAssist^TM Program Implementation

INTERVENTIONS:
Other: Senior PharmAssist^TM Program Implementation — Representatives from three diverse communities will participate in co-design workshops to refine the Senior PharmAssistTM (SPA) implementation toolkit, which will then be delivered to agency staff from these partnering communities through a series of learning collaborative sessions to facilitate implementation of SPA core components in each community.
  Community champions will be trained to deliver a community-based program to deliver the core components of SPA:
  1. Medication Therapy Management (MTM);
  2. Medication co-payment assistance;
  3. Tailored community referrals; and
  4. Medicare insurance counseling

SUMMARY:
This project aims to evaluate the scalability of an established, evidence-based, multi-component intervention, Senior PharmAssist^TM (SPA), designed to improve function and quality of life of older adults with limited incomes. The investigators propose to refine existing SPA replication materials such as community readiness assessments, educational tools to facilitate implementation of care processes, and data collection tools for quality improvement with input from community stakeholders interested in implementation of the SPA intervention. After gathering feedback from key stakeholders in 3 diverse communities in North Carolina, and refining tools accordingly, SPA staff will then provide technical assistance to support implementation in these communities, using the Institute for Healthcare Improvement learning collaborative approach, to facilitate community agency staff implementation of the SPA core components with racially diverse older adults with limited incomes using small scale tests of change with feedback.

The investigators will collect data from key stakeholders including older adults, community volunteers, and agency staff regarding facilitators and barriers to implementation of SPA, and obtain aggregate data regarding older adult participants served, including demographics, participant satisfaction, and self-rated health. Data will be analyzed using a multiple case study design that incorporates both qualitative data on barriers and facilitators, as well as aggregated data on older adults enrolled in community programs.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 or older
* Currently or soon to be enrolled in Medicare
* Income is at or below 200% of Poverty Line
* Lives in one of 3 targeted communities learning to implement the Senior PharmAssist^TM core services
* Seeks assistance with medications, Medicare counseling, or tailored referrals from agencies participating in Senior PharmAssist^TM learning collaborative

Exclusion Criteria:

None

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor McConnell, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Communities Adopting Senior PharmAssist Implementation Toolkit: Three communities will commit to learning how to implement the evidence-based, multi-component intervention, Senior PharmAssistTM (SPA), designed to improve function and quality of life of older adults with limited incomes using the SPA toolkit.
  The toolkit, co-developed with community leaders, will help to create a community model for implementation that addresses equitable access to medications, medication management, and community supports that promote physical function and healthy aging in place.
  Senior PharmAssist^TM Program Implementation: Representatives from three diverse communities will participate in co-design workshops to refine the Senior PharmAssistTM (SPA) implementation toolkit, which will then be delivered to agency staff from these partnering communities through a series of learning collaborative sessions to facilitate implementation of SPA core components in each community.
  Community champions will be trained to deliver a community-based program to deliver the core components of SPA:
  1. Medication Therapy Management (MTM);
  2. Medication co-payment assistance;
  3. Tailored community referrals; and
  4. Medicare insurance counseling
Period: Overall Study
Arm/Group | Communities Adopting Senior PharmAssist Implementation Toolkit
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Communities Adopting Senior PharmAssist Implementation Toolkit
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Older Adults Seeking Service Who Received All 4 Components of Senior PharmAssist Intervention
Time Frame: 13 months post-completion of learning collaborative
Measure: Count of Participants; unit: Participants
Arm/Group | Communities Adopting Senior PharmAssist Implementation Toolkit
Number analyzed (Participants) | 7
Participants | 0

2. Secondary Outcome: Percentage of Older Adults Receiving Medication Therapy Management
Time Frame: 13 months post-completion of learning collaborative
Measure: Number; unit: percentage of participants
Arm/Group | Communities Adopting Senior PharmAssist Implementation Toolkit
Number analyzed (Participants) | 7
percentage of participants | 100

3. Secondary Outcome: Percentage of Older Adults Receiving Medication Co-pay Assistance
Time Frame: 13 months post-completion of learning collaborative
Measure: Number; unit: percentage of participants
Arm/Group | Communities Adopting Senior PharmAssist Implementation Toolkit
Number analyzed (Participants) | 7
percentage of participants | 28.57

4. Secondary Outcome: Percentage of Older Adults Receiving at Least One Tailored Community Referral
Time Frame: 13 months post-completion of learning collaborative
Measure: Number; unit: percentage of participants
Arm/Group | Communities Adopting Senior PharmAssist Implementation Toolkit
Number analyzed (Participants) | 7
percentage of participants | 42.86

5. Secondary Outcome: Percentage of Older Adults Receiving Medicare Counseling
Time Frame: 13 months post-completion of learning collaborative
Measure: Number; unit: percentage of participants
Arm/Group | Communities Adopting Senior PharmAssist Implementation Toolkit
Number analyzed (Participants) | 7
percentage of participants | 71.43

6. Other Pre Specified Outcome: Change in Self-rated Health
Description: Change from baseline in proportion of participants who rate their health as good to excellent.
  Scale of rating ranges from 1 = poor, 2 = fair, 3 = good, 4 = very good, 5 = excellent.
Time Frame: Baseline, 13 months post-completion of learning collaborative
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 13 months post-completion of learning collaborative
Arm/Group | Communities Adopting Senior PharmAssist Implementation Toolkit
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/50/NCT05278650/Prot_SAP_001.pdf
  • Informed Consent Form (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT05278650/ICF_000.pdf